CLINICAL TRIAL: NCT05411354
Title: Analyzing Clinical Trial Experiences of Prostate Cancer Patients To Determine How Trial Attributes Affect Completion Rates For Specific Demographic Groups
Brief Title: Analyzing Clinical Trial Experiences of Prostate Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 585375c1448bfa3494298bdd794080
Record Dates: First submitted 2022-06-05; First posted 2022-06-09 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate; Prostate Clinical Trials
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in clinical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the participation or completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of Prostate Cancer patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might shed insights for the sake of future Prostate Cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with Prostate Cancer as identified by imaging
* Patient has self-identified as planning to enroll in an interventional clinical trial for Prostate Cancer
* Patient is at least 18 years of age

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient has a ECOG score of 4

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer patients who are actively considering enrolling in an interventional clinical trial to treat their Prostate Cancer, but have yet to complete randomization and enrollment.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a Prostate Cancer Clinical Trial | 3 months
Number of patients who remain in Prostate Cancer clinical trial until completion of clinical trial | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Science Inc
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McKay RR, Gold T, Zarif JC, Chowdhury-Paulino IM, Friedant A, Gerke T, Grant M, Hawthorne K, Heath E, Huang FW, Jackson MD, Mahal B, Ogbeide O, Paich K, Ragin C, Rencsok EM, Simmons S, Yates C, Vinson J, Kantoff PW, George DJ, Mucci LA. Tackling Diversity in Prostate Cancer Clinical Trials: A Report From the Diversity Working Group of the IRONMAN Registry. JCO Glob Oncol. 2021 Apr;7:495-505. doi: 10.1200/GO.20.00571. PMID 33835826
- [Background] Rencsok EM, Bazzi LA, McKay RR, Huang FW, Friedant A, Vinson J, Peisch S, Zarif JC, Simmons S, Hawthorne K, Villanti P, Kantoff PW, Heath E, George DJ, Mucci LA. Diversity of Enrollment in Prostate Cancer Clinical Trials: Current Status and Future Directions. Cancer Epidemiol Biomarkers Prev. 2020 Jul;29(7):1374-1380. doi: 10.1158/1055-9965.EPI-19-1616. Epub 2020 Jun 5. PMID 32503813

DOCUMENTS (1):
  • Informed Consent Form (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT05411354/ICF_000.pdf